CLINICAL TRIAL: NCT02655094
Title: Unilateral Pulmonary Edema After Minimal-invasive Mitral Valve Surgery: a Retrospective Single Center Observation
Brief Title: Unilateral Pulmonary Edema After Minimal-invasive Mitral Valve Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PD Dr., University Hospital Schleswig-Holstein
Other Study IDs: IN-MIC-01
Record Dates: First submitted 2015-12-05; First posted 2016-01-13 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Edema
Keywords: minimal-invasive surgery, mitral valve
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Unilateral pulmonary edema after minimal-invasive mitral valve surgery is a rare but in some cases severe complications, sometimes causing extracorporeal life support. The investigators have observed over several years 5 cases of instantaneous postoperative severe pulmonary edema. This is a retrospective analysis of over 200 minimal-invasive mitral valve surgery procedure.

DETAILED DESCRIPTION:
Unilateral pulmonary edema after minimal-invasive mitral valve surgery is a rare but in some cases severe complications, sometimes causing extracorporeal life support. The investigators have observed over several years 5 cases of instantaneous postoperative severe pulmonary edema. After having studied the available literature on this particular topic the investigators have decided to prepare a retrospective analysis of over 200 minimal-invasive mitral valve surgery procedure focusing on radiological and clinical signs of unilateral pulmonary edema.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age

Exclusion Criteria:

* urgent surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collective of patients with relevant mitral valve disease scheduled for minimal-invasive mitral valve repair or replacement
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Unilateral right sided pulmonary edema or congestion after surgery | Postoperatively within the first 12h after admission to intensive care unit
  retrospective analysis using the electronic and the paper-based patient specific database

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, PD Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renner J, Lorenzen U, Borzikowsky C, Schoeneich F, Cremer J, Haneya A, Hensler J, Panholzer B, Huenges K, Broch O. Unilateral pulmonary oedema after minimally invasive mitral valve surgery: a single-centre experience. Eur J Cardiothorac Surg. 2018 Apr 1;53(4):764-770. doi: 10.1093/ejcts/ezx399. PMID 29186375